CLINICAL TRIAL: NCT02277665
Title: Randomized Trial Evaluating Treatment for Cannabis Use Disorders Among Those Who Use Tobacco
Brief Title: Clinical Trial Tobacco Marijuana
Acronym: RCTTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alan J. Budney, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00028307 D14233; 5R01DA032243 (NIH)
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Cannabis Use Disorder; Tobacco Use Disorder
Keywords: Cannabis Use Disorder; Tobacco Use; Treatment
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use | interventions — Cognitive Behavioral Therapy; Behavior Therapy; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CUD Treatment Only (Active Comparator): 12 Week Behavioral Treatment that included weekly computer-assisted counseling and contingency management for CUD
  Interventions: Behavioral: CUD Treatment
- CUD and Tobacco Treatment (Experimental): 12 Week Behavioral Treatment that included weekly computer-assisted counseling and contingency management for CUD, and behavioral counseling and nicotine replacement therapy (NRT) for tobacco
  Interventions: Behavioral: CUD Treatment; Behavioral: Tobacco Treatment

INTERVENTIONS:
Behavioral: CUD Treatment
  Other Names: Cognitive Behavioral Therapy and Contingency Management
Behavioral: Tobacco Treatment
  Other Names: Behavioral Counseling plus NRT
  Arms: CUD and Tobacco Treatment

SUMMARY:
Approximately 50% of persons seeking treatment for cannabis-use disorders (CUDs) regularly smoke tobacco. Combining tobacco with cannabis has become a common method of smoking cannabis. Similarities of use, and using together, can make quitting difficult. Stopping tobacco simultaneously with cannabis may be beneficial. Little scientific information currently addresses how to best target tobacco smoking during treatment for CUDs. Our long-term goal is to develop an effective protocol for intervening in tobacco smoking without changing cannabis outcomes.

This protocol reflects the planned Stage 1, proof-of-concept study that will compare a combined cannabis and tobacco intervention to one that targets CUD only. Hypotheses assert that the intervention (1) will be accepted by the majority of eligible participants (2) will result in more tobacco quit attempts and rates than the CUD-only treatment; and (3) will not adversely affect cannabis outcomes. Last, the project will evaluate the potential of specific moderators of outcomes to predict outcomes and inform subsequent treatment development efforts. If the hypotheses were confirmed, dissemination of this protocol would reduce adverse psychosocial and health consequences of tobacco or cannabis dependence. Findings will inform future development of prevention and intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals must be 18 years or older
2. Individuals must meet criteria for the current Diagnostic and Statistical Manual -IV diagnosis of cannabis abuse or dependence, report use of cannabis on at least 45 of the previous 90 days, and report regular use of tobacco cigarettes or report that their primary administration of cannabis is via blunts or spliffs
3. Individual must indicate that they have at least some interest in quitting tobacco in the next 6 months (rating of 2 or more on a 5-point interest scale)

Exclusion Criteria:

1. Current dependence on alcohol or any drug other than tobacco and cannabis
2. Use of non-tobacco nicotine
3. Current participation in structured treatment for substance abuse
4. Severe psychological distress (e.g., active suicidal plans, psychosis, debilitating panic disorder)
5. Report of a condition that requires seeing a physician before using NRT (e.g., pregnancy or recent heart attack); note: if a participant's physician approves taking NRT, we will consider enrolling them
6. Legal status that would interfere with participation
7. Living with someone currently enrolled in the project
8. Not being fluent in English
9. Not living within 45 miles of the research site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Budney, Ph.D, Principal Investigator — Dartmouth-Hitchcock Medical Center; Denise Walker, Ph.D, Principal Investigator — University of Washington School of Social Work
Locations (3):
- United States (3):
  - Geisel School of Medicine at Dartmouth; State Building Site, Concord, New Hampshire
  - Geisel School of Medicine at Dartmouth; Rivermill Complex Site, Lebanon, New Hampshire
  - University of Washington School of Social Work, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between 12/2014 to 09/2016 at Dartmouth College and the University of Washington. Participants were recruited from ads posted online (Craigslist, Facebook), in newspapers, on radio, community posters, and notices to service agencies. All activities occurred at stand-alone, University associated research clinics.
Pre-assignment Details: All those who enrolled were assigned to a treatment condition
Groups:
- CUD Treatment Only: 12 Week Behavioral Treatment that included weekly computer-assisted counseling and contingency management for CUD
  CUD Treatment
- CUD and Tobacco Treatment: 12 Week Behavioral Treatment that included weekly computer-assisted counseling and contingency management for CUD, and behavioral counseling and nicotine replacement therapy (NRT) for tobacco
  CUD Treatment
  Tobacco Treatment
Period: Overall Study
Arm/Group | CUD Treatment Only | CUD and Tobacco Treatment
Started | 33 | 34
Completed | 33 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CUD Treatment Only | CUD and Tobacco Treatment | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (12.2) | 31.7 (11.2) | 34.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 25 | 23 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 22 | 21 | 43
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Tobacco Quit Attempts
Description: Percent of Participants who made at least one tobacco quit attempt
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | CUD Treatment Only | CUD and Tobacco Treatment
Number analyzed (Participants) | 33 | 34
Participants | 13 | 17
Statistical Analysis 1: Comparison: CUD Treatment Only vs CUD and Tobacco Treatment; Test type: Superiority — Chi-square; p = 0.33, Chi-squared; Odds Ratio (OR) = 0.56, 95% CI 2-sided [.17 to 1.82]

2. Primary Outcome: Tobacco Abstinence
Description: the percent of participants who achieve sustained tobacco abstinence, which reflects biologically-verified abstinence during weeks 5-12
Time Frame: Weeks 9-12
Measure: Count of Participants; unit: Participants
Arm/Group | CUD Treatment Only | CUD and Tobacco Treatment
Number analyzed (Participants) | 33 | 34
Participants | 1 | 2
Statistical Analysis 1: Comparison: CUD Treatment Only vs CUD and Tobacco Treatment; Test type: Other; p = 0.57, Chi-squared; Odds Ratio (OR) = 0.32

3. Primary Outcome: Cannabis Abstinence
Description: number of participants who achieved at least one week of documented cannabis abstinence during treatment
Time Frame: Weeks 1-12
Measure: Count of Participants; unit: Participants
Arm/Group | CUD Treatment Only | CUD and Tobacco Treatment
Number analyzed (Participants) | 33 | 34
Participants | 12 | 7
Statistical Analysis 1: Comparison: CUD Treatment Only vs CUD and Tobacco Treatment; Test type: Other; p = 0.16, Chi-squared; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.15 to 1.35]

4. Primary Outcome: Weeks of Continuous Cannabis Abstinence
Description: Weeks of Continuous Cannabis Abstinence among those achieving at least one week of abstinence
Time Frame: Weeks 1-12
Population: All participants
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | CUD Treatment Only | CUD and Tobacco Treatment
Number analyzed (Participants) | 33 | 34
weeks | 6.1 (3.7) | 5.9 (4.0)
Statistical Analysis 1: Comparison: CUD Treatment Only vs CUD and Tobacco Treatment; Test type: Superiority; p = 0.87, Chi-squared; Means Ratio = 0.97, 95% CI 2-sided [0.66 to 1.42]

5. Primary Outcome: Treatment Attendance
Description: Attendance operationalized as the number of clinic visits (urine specimens provided)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: visits
Groups:
- CUD Treatment: Received CUD treatment and delayed Tobacco Intervention
- CUD Treatment and Tobacco Intervention: Received CUD treatment and Tobacco Intervention simultaneously
Arm/Group | CUD Treatment | CUD Treatment and Tobacco Intervention
Number analyzed (Participants) | 33 | 34
visits | 11.3 (9.0) | 9.7 (8.9)
Statistical Analysis 1: Comparison: CUD Treatment vs CUD Treatment and Tobacco Intervention; Test type: Superiority; p = 0.46, t-test, 2 sided

6. Primary Outcome: Initiation of Nicotine Replacement Therapy (NRT)
Description: # of participants who initiated NRT during the 24 week study period
Time Frame: 24 weeks
Population: All participants included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | CUD Treatment | CUD Treatment and Tobacco Intervention
Number analyzed (Participants) | 33 | 34
Participants | 6 | 14
Statistical Analysis 1: Comparison: CUD Treatment vs CUD Treatment and Tobacco Intervention; Test type: Superiority; p = 0.04, Chi-squared

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | CUD Treatment Only | CUD and Tobacco Treatment
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 3/33 | 5/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CUD Treatment Only (N=33) | CUD and Tobacco Treatment (N=34)
pruritus (Endocrine disorders) | 3 (3) | 5 (5)

LIMITATIONS AND CAVEATS:
Enrollment did not meet planned target numbers, limiting the power to detect differences between conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT02277665/Prot_SAP_000.pdf